CLINICAL TRIAL: NCT02072174
Title: International Multicenter Double-blind Placebo-controlled Randomized Parallel Group Clinical Trial of Efficacy of Anaferon for Children in the Treatment of Influenza and Acute Respiratory Viral Infections in Children
Brief Title: Efficacy of Anaferon for Children in the Treatment of Influenza and Acute Respiratory Viral Infections in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-AD-004
Record Dates: First submitted 2014-02-14; First posted 2014-02-26 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Influenza and Acute Respiratory Viral Infections
MeSH Terms: conditions — Influenza, Human | interventions — anaferon; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaferon for Children (Experimental): On day 1, five tablets are taken in the first 2 hours (one tablet every 30 min), followed by three more tablets regularly spaced during the rest of the day. From day 2 through 5, one tablet is administered three times daily.
  Interventions: Drug: Anaferon for Children
- Placebo (Placebo Comparator): On day 1, five tablets are taken in the first 2 hours (one tablet every 30 min), followed by three more tablets regularly spaced during the rest of the day. From day 2 through 5, one tablet is administered three times daily.
  Interventions: Drug: Anaferon for Children

INTERVENTIONS:
Drug: Anaferon for Children — Anaferon for children: For oral use.
  Other Names: Anaferon for Children in tablets

SUMMARY:
The purpose of this study is:

• To obtain additional data on therapeutic efficacy of Anaferon for children in the treatment of influenza and acute respiratory viral infections in children

DETAILED DESCRIPTION:
The study will enroll outpatient subjects of both sexes aged 3-12 years with clinical manifestations of influenza/Acute Respiratory Viral Infections (ARVI), including fever

≥ 38.0°С having an appointment with a doctor within the first day after the illness onset.

Тhe physician will collect medical history information, perform an objective examination, record the concomitant therapy, and obtain nasal swab specimens for a rapid diagnostic influenza test. If the swab is positive, the doctor shall obtain swab specimens from the nasal cavity and oropharynx (nasopharyngeal swab) for a subsequent real time reverse transcription-polymerase chain reaction (RT-PCR) to determine the viral load of influenza A and/or B virus. If the swab is negative for influenza the doctor shall collect a nasopharyngeal swab for a subsequent PCR test for other respiratory viruses.

If inclusion criteria are met and exclusion criteria are absent at visit 1 (Day 1), the patient will be enrolled in the trial and randomized into one of the two groups: group 1 patients will take Anaferon for children following a 5-day regimen; group 2 patients will receive Placebo using the Anaferon for children 5-day regimen. The parent/adopter of patient will receive a diary where they should record the child's axillary temperature data in the morning and evening, and score the severity of symptoms.

The subject will be monitored for 14 days (screening, randomization - 1 day, treatment - 5 days, follow-up - 1 day; late-scheduled phone "visit" - day 14).

At Visits 2-4, the physician will document objective examination data; obtain nasopharyngeal swabs from subjects with positive influenza tests for subsequent RT-PCR to determine the viral load and its reduction in the course of treatment; monitor the prescribed and concomitant therapy, and check the patient's diary data. The phone "visit" will be made to elicit information from the parents regarding the patient's general health, presence/absence of secondary bacterial/viral complications, and use of antibacterial drugs.

Interim statistical analysis is stipulated by the study protocol. Interim analysis will be performed using the data obtained from the examination and treatment of the protocol-defined number of patients who completed the study. Based on the expected effect, the minimum required Particular Per Protocol (pPP) sample size will be 254 patients (127 subjects in each group - Anaferon for children and Placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged 3-12 years inclusively.
2. Diagnosis of influenza/ARVI according to physician's examination: body temperature ≥ 38.0°C at the time of examination + symptom score ≥ 4 (at least 1 systemic symptom ≥2 and 1 nasal/throat/chest symptom ≥2 or several symptoms ≥ 1 score).
3. The first 24 hours from the beginning of manifestations of influenza/ARVI.
4. The possibility to start therapy within 24 hours from the first symptoms of ARVI.
5. Availability of a patient information sheet (Informed Consent form) for parents/adoptive parents for participation in the study signed by one of the parents/adoptive parents.

Exclusion Criteria:

1. Suspected pneumonia, bacterial infection or severe disease requiring antibacterial products (including sulfanilamides) starting from the first day of the disease.
2. Clinical symptoms of severe influenza/ARVI requiring hospitalization.
3. Suspected initial manifestations of the diseases having the symptoms similar to the ones of influenza/ARVI (other infectious diseases, influenza-like syndrome at debut of systemic connective tissue diseases, oncohematological and other diseases).
4. Medical history of primary and secondary immunodeficiencies: а) lymphoid system immunodeficiencies (Т-cell and/or B-cell, immunodeficiencies with predominant antibody deficiency); b) phagocytic deficiencies; c) complement factor deficiency; d) combined immunodeficiencies including AIDS secondary to HIV-infection; toxic, autoimmune, infectious, radiation panleukopenic syndrome; systemic lymphocytopenic syndrome; polyclonal lymphocytic activation syndrome; postsplenectomic syndrome; congenital asplenia; immune complex pathological syndrome associated with infectious, autoimmune and allergic diseases.
5. Medical history of sarcoidosis.
6. Oncology.
7. Exacerbation or decompensation of chronic diseases affecting ability to participate in the clinical study.
8. Medical history of polyvalent allergy.
9. Allergy/intolerance to any of the components of medications used in the treatment.
10. Malabsorption syndrome, including congenital or acquired lactase or other disaccharidase deficiency, galactosemia.
11. Intake of medicines listed in the section "Prohibited concomitant therapy" within 1 month prior to the inclusion in the study.
12. Drug addiction, alcohol consumption at more than 2 alcohol units per day by the subject's parents/adoptive parents.
13. Mental diseases of the subject, parents/adoptive parents.
14. Subjects whose parents/adoptive parents, according to the investigator's point of view, will not follow the observation requirements during the study or study product dosing regimen.
15. Participation in other clinical studies within 3 months prior to the inclusion in the study.
16. Parent/adoptive parent of the subject is related to the investigator team of medical facility directly involved in the study or is a close relative of the investigator. Close relatives include spouse, parents, children or brothers (sisters) regardless of whether they are biological or adoptive ones.
17. Parent/adoptive parent of the subject is working in OOO "NPF "Materia Medica Holding", i.e. is the company official, temporary contract worker or an appointed official responsible for the study or their close relatives.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 569 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Andrianova, Professor, Study Director — Materia Medica Holding
Locations (27):
- Belarus (3):
  - City Child Health Clinical Polyclinic №13, Minsk
  - Municipal Health Care Institution "City Child Health Clinical Polyclinic №10", Minsk
  - City Child Health Clinical Polyclinic №17, Minsk
- Russia (22):
  - Clinic of State Budgetary Institution "Research Institute of nutrition" of the Russian Academy of Medical Sciences, Moscow
  - Russian National Research Medical University named after N.I. Pirogov, Moscow
  - Russian National Research Medical University, Moscow
  - Russian National Research Pirogov Medical University, Moscow
  - State Educational Institution of Higher Professional Education "Moscow State Medical Academy named after I.M. Sechenov", Moscow
  - State Budgetary Institution of Health, "Children's City Hospital № 9 named after G.N. Speranskii", Moscow
  - State Budgetary Educational Institution of Additional Professional Education "Russian Russian Medical Academy of Postgraduate Education" of Ministry of Health of Russian Federation, Moscow
  - State Budgetary Educational Institution of Higher Professional Education " Nizhny Novgorod State Medical Academy" of Ministry of Health of Russian Federation, Nizhny Novgorod
  - State Budgetary Educational Institution of Higher Professional Education ''Novosibirsk State Medical University'' of Ministry of Health of Russian Federation, Novosibirsk
  - Municipal Health Care Institution "City Child Health Clinical Polyclinic №5", Perm
  - State Budgetary Educational Institution of Higher Professional Education "Rostov State Medical University", Rostov-on-Don
  - St. Petersburg State Budgetary Health Care Institution "Сity Polyclinic №44", Saint Petersburg
  - St. Petersburg State health institution " City Child Health Polyclinic № 45", Saint Petersburg
  - State Budgetary Educational Institution of Higher Professional Education "St. Petersburg State Pediatric Medical Academy" of Ministry of Health of Russian Federation, Saint Petersburg
  - Limited Liability Company "Alliance Biomedical-Russian group", Saint Petersburg
  - Co.Ltd "Clinic Allergomed", Saint Petersburg
  - State Health Care Institution "Child Health City Hospital №22", Saint Petersburg
  - Bashkir State Medical University of Ministry of Health of Russian Federation, Ufa
  - State Budgetary Educational Institution of Higher Professional Education " Yaroslavl State Medical Academy" of Ministry of Health of Russian Federation, Yaroslavl
  - State Budgetary Educational Institution of Higher Professional Education "Yaroslavl State Medical Academy", Yaroslavl
  - State Budgetary Educational Institution of Higher Professional Education "Yaroslavl State Medical Academy, Yaroslavl
  - Yaroslavl State Medical Academy, Yaroslavl
- Ukraine (2):
  - Vinnytsya M.I. Pyrogov National Medical University, Vinnytsia
  - Public institution "Zaporizhzhya city multidisciplinary children's hospital №5", Zaporozh’ye

RESULTS

PARTICIPANT FLOW:
Groups:
- Anaferon for Children: Anaferon for Children: 1 tablet per 1 intake. On the first day of treatment: the first 2 hours of 1 tablet every 30 minutes, then, during the first day, 3 more times at regular intervals. From the second to the fifth day: 1 tablet 3 times a day. The drug is taken out of the reception of food (in the interval between meals or 15-30 minutes before eating), should be kept in your mouth, not swallowed, until it is dissolved completely.
- Placebo: Placebo: 1 tablet per 1 intake. On the first day of treatment: the first 2 hours of 1 tablet every 30 minutes, then, during the first day, 3 more times at regular intervals. From the second to the fifth day: 1 tablet 3 times a day. The drug is taken out of the reception of food (in the interval between meals or 15-30 minutes before eating), should be kept in your mouth, not swallowed, until it is dissolved completely.
Period: Overall Study
Arm/Group | Anaferon for Children | Placebo
Started | 290 | 279
Completed | 258 | 240
Not Completed | 32 | 39
Not completed — Did Not Meet In-/Exclusion Criteria | 14 | 15
Not completed — Protocol Violation | 16 | 23
Not completed — Physician Decision | 0 | 1
Not completed — Non-compliance with protocol requirement | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaferon for Children | Placebo | Total
Number analyzed (Participants) | 258 | 240 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.8 (2.7) | 6.7 (2.7) | 6.7 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 115 | 233
  Male | 140 | 125 | 265
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Count of Participants [Count of Participants; unit: Participants] | 258 | 240 | 498

OUTCOME MEASURES:

1. Primary Outcome: Average Illness Duration
Description: Disease duration is assessed until recovery or significant improvement. Average illness duration is defined as the interval between the start of the trial treatment and the start of the first 24-hour period in which the non-specific symptoms and nasal/ throat/ chest symptoms improve to "absent" or "mild" (Total Symptom Score of severity had decreased to ≤2 points) and body temperature returns to 37.2°C or below.
  Based on patient diary data.
Time Frame: From the time of randomization until the time of recovery/improvement (days 1-14)
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 258 | 240
days | 4.6 (1.4) | 4.9 (1.3)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.0242, Kruskal-Wallis

2. Secondary Outcome: Percentage of Patients With Recovery/Improvement in Health
Description: Based on Days 2, 3, 4 and 5 of observation treatment (according to the patient's diary), on days 3 and 5 of therapy (according to physician's objective examination).
Time Frame: on days 2, 3, 4 and 5 of the treatment
Population: Per Protocol set
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 258 | 240
Participants
  Day 2 (patient diary data) | 1 | 1
  Day 3 (patient diary data) | 25 | 11
  Day 4 (patient diary data) | 61 | 40
  Day 5 (patient diary data) | 107 | 84
  Day 3 (physician's examination) | 31 | 16
  Day 5 (physician's examination) | 116 | 90
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; patient diary data; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Anaferon for Children vs Placebo; doctor's examination data; Test type: Superiority; p = 0.0127, Cochran-Mantel-Haenszel

3. Secondary Outcome: Changes in Body Temperature
Description: Changes in Body Temperature Based on Patient Diary Data
Time Frame: baseline and days 2, 3, 4 and 5 of observation treatment
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 258 | 240
°C
  Day 1 | 38.5 (0.4) | 38.5 (0.4)
  Day 2 | 38.0 (0.8) | 38.2 (0.8)
  Day 3 | 37.4 (0.8) | 37.5 (0.8)
  Day 4 | 37.0 (0.6) | 37.1 (0.7)
  Day 5 | 36.8 (0.4) | 36.9 (0.4)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.0394, Mixed Models Analysis — The p-value associated with "treatment" factor of variable on day 2, 3, 4 and 5 between Anaferon for Children and Placebo. Model includes treatment, visit, treatment*visit interaction, Day 1 covariate. Treatment*visit interaction p-value is 0.3220
Statistical Analysis 2: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.3220, Mixed Models Analysis — The p-value associated with "treatment*visit" interaction factor of variable on day 2, 3, 4 and 5 between Anaferon for Children and Placebo. Model includes treatment, visit, treatment*visit interaction, Day 1 covariate

4. Secondary Outcome: Percentage of Patients With Normal Body Temperature (≤37.0ºС)
Description: Based on the patient diary data. Axillary temperature (morning and evening) decline to or below 37.0 ºС.
Time Frame: on days 2, 3, 4 and 5 of observation treatment
Population: Per Protocol set
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 258 | 240
Participants
  Day 2 (patient diary data) | 31 | 23
  Day 3 (patient diary data) | 104 | 76
  Day 4 (patient diary data) | 167 | 139
  Day 5 (patient diary data) | 219 | 196
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.0043, Cochran-Mantel-Haenszel

5. Secondary Outcome: Severity of Clinical Manifestations of Influenza / Acute Respiratory Viral Infection by Total Symptom Score.
Description: Total Symptom Score is based on the severity of each Influenza / Acute Respiratory Viral Infection symptom.
  Total Symptom Score includes 13 symptoms: body temperature, non-specific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness), nasal/throat/chest symptoms.
  The severity of non-specific and nasal/throat/chest symptom is scored on a symptom severity scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms).
  Minimum score=0; maximum score=39. The severity of symptoms is recorded by the doctors on the case record form on days 3, 5 and by parents/adopter on a diary card twice a day on days 2-6.
Time Frame: on days 2-6 of observation treatment
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 258 | 240
score on a scale
  Day 2 (patient diary data) | 10.0 (5.3) | 11.0 (5.1)
  Day 3 (patient diary data) | 7.0 (4.8) | 8.1 (4.8)
  Day 4 (patient diary data) | 5.0 (3.8) | 5.5 (3.8)
  Day 5 (patient diary data) | 3.3 (2.9) | 3.8 (3.1)
  Day 3 (physician's examination) | 7.0 (4.6) | 8.1 (4.8)
  Day 5 (physician's examination) | 3.5 (3.0) | 3.9 (3.0)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Day 2 (patient diary data); Test type: Superiority; p = 0.0104, Kruskal-Wallis — p-value not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Anaferon for Children vs Placebo; Day 3 (patient diary data); Test type: Superiority; p = 0.0041, Kruskal-Wallis — p-value not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Anaferon for Children vs Placebo; Day 4 (patient diary data); Test type: Superiority; p = 0.0484, Kruskal-Wallis — p-value not adjusted for multiple comparisons
Statistical Analysis 4: Comparison: Anaferon for Children vs Placebo; Day 5 (patient diary data); Test type: Superiority; p = 0.0603, Kruskal-Wallis — p-value not adjusted for multiple comparisons
Statistical Analysis 5: Comparison: Anaferon for Children vs Placebo; Day 3 (doctor's examination); Test type: Superiority; p = 0.0056, Kruskal-Wallis — p-value not adjusted for multiple comparisons
Statistical Analysis 6: Comparison: Anaferon for Children vs Placebo; Day 5 (doctor's examination); Test type: Superiority; p = 0.0994, Kruskal-Wallis — p-value not adjusted for multiple comparisons

6. Secondary Outcome: Assessment of the Severity of Influenza Virus / Acute Respiratory Viral Infection Using the "Area Under the Curve" for an Overall Symptom Assessment
Description: Total Symptom Score is based on the severity of each disease symptom. The TSS includes 13 symptoms: body temperature/fever, non-specific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness), nasal/throat/chest symptoms (runny nose, nasal congestion, sneezing, sore throat, hoarseness, cough, chest pain/tightness of the chest).
  Minimum score=0; maximum score=39. The area under the curve 1 = on days 1, 3, 5 and 7 on the results of doctor's examination The area under the curve 2 = based on days 1-7 on the patient diary data
Time Frame: on days 1-7 of observation (based on days 1-7 on the patient diary data; on days 1, 3, 5 and 7 of observation - according to physician's objective examination)
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: score*day
Groups:
- Anaferon for Children: Anaferon for children: Anaferon for children: 1 tablet per 1 intake. On the first day of treatment: the first 2 hours of 1 tablet every 30 minutes, then, during the first day, 3 more times at regular intervals. From the second to the fifth day: 1 tablet 3 times a day. The drug is taken out of the reception of food (in the interval between meals or 15-30 minutes before eating), should be kept in your mouth, not swallowed, until it is dissolved completely.
- Placebo: Placebo: Placebo: 1 tablet per 1 intake. On the first day of treatment: the first 2 hours of 1 tablet every 30 minutes, then, during the first day, 3 more times at regular intervals. From the second to the fifth day: 1 tablet 3 times a day. The drug is taken out of the reception of food (in the interval between meals or 15-30 minutes before eating), should be kept in your mouth, not swallowed, until it is dissolved completely.
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 258 | 240
score*day
  Days 1-7 (patient diary data) | 34.4 (18.8) | 38.2 (18.5)
  Days 1, 3, 5 and 7 (physician's examination) | 17.6 (8.9) | 19.3 (8.9)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Days 1-7 (patient diary data); Test type: Superiority; p = 0.0084, Kruskal-Wallis
Statistical Analysis 2: Comparison: Anaferon for Children vs Placebo; Days 1, 3, 5 and 7 (doctor's examination); Test type: Superiority; p = 0.0233, Kruskal-Wallis

7. Secondary Outcome: Number of Intakes of Antipyretics
Description: Number of Intakes of Antipyretics based on patient diary data
Time Frame: on days 1-5 of therapy
Population: Per Protocol set
Measure: Mean (Standard Deviation); unit: Number of intakes
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 258 | 240
Number of intakes
  Day 1 | 1.2 (0.9) | 1.3 (1.0)
  Day 2 | 0.7 (1.0) | 0.9 (1.1)
  Day 3 | 0.3 (0.6) | 0.4 (0.8)
  Day 4 | 0.1 (0.4) | 0.1 (0.5)
  Day 5 | 0.0 (0.2) | 0.1 (0.4)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.0721, Mixed Models Analysis

8. Secondary Outcome: Change in Viral Load During the Treatment and Follow-up Periods
Description: Viral load is evaluated in subjects with positive influenza A and B tests. Virus load [log10 copies influenza А/В RNA per 1 mL] in nasal and pharyngeal swabs is determined using real-time PCR on days 1, 3, 5 and 7.
Time Frame: on days 1, 3, 5, 7 of observation treatment
Population: Viral load is evaluated in subjects with positive influenza A and B tests.
Measure: Mean (Standard Deviation); unit: log10 copies influenza А/В RNA per 1 mL
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 49 | 51
log10 copies influenza А/В RNA per 1 mL
  Day 1 | 5.7 (1.1) | 5.6 (1.3)
  Day 3 | 4.1 (2.2) | 4.8 (1.3)
  Day 5 | 3.1 (2.3) | 4.4 (1.3)
  Day 7 | 2.1 (2.4) | 4.0 (1.5)
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.0001, Mixed Models Analysis

9. Secondary Outcome: Percentage of Patients With Exacerbation of the Disease Course
Description: The development of disease complications requiring antibiotics drugs or hospitalization
Time Frame: 14 days of observation treatment
Population: Per Protocol set
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 258 | 240
Participants | 7 | 11
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.3383, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered during 14 days (during the treatment and follow-up periods ).
Description: Adverse/Serious adverse events were registered in patients of the Safety population (n=569)
Arm/Group | Anaferon for Children | Placebo
All-Cause Mortality (participants affected / at risk) | 0/290 | 0/279
Serious Adverse Events (participants affected / at risk) | 1/290 | 1/279
Other Adverse Events (participants affected / at risk) | 26/290 | 30/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaferon for Children (N=290) | Placebo (N=279)
Influenza (Infections and infestations) | 1 (1) | 1 (1) — Hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaferon for Children (N=290) | Placebo (N=279)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Adenoiditis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3) | 4 (4)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (3)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysbacteriosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Otitis media acute (Infections and infestations) | 4 (4) | 5 (5)
Otosalpingitis (Infections and infestations) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT02072174/Prot_SAP_000.pdf